CLINICAL TRIAL: NCT06506643
Title: A Phase I/II Open-label Multicenter Dose Escalation and Dose Expansion Study to Evaluate the Safety and Efficacy of KLS-1 as Monotherapy in Patients With Malignant Neoplasms
Brief Title: Safety and Efficacy of KLS-1 Monotherapy in Malignant Neoplasms
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vector Vitale LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VV022-02
Record Dates: First submitted 2024-06-07; First posted 2024-07-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: CLL; Solid Tumor, Adult
Keywords: malignant melanoma; prostate cancer; pancreatic cancer; CLL; chronic lymphocytic leukemia; Zn; Zinc; KLS-1; Malignant Neoplasms; Neoplasms; Metastatic Tumors; Zinc Aspartate
MeSH Terms: conditions — Melanoma; Prostatic Neoplasms; Pancreatic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Phase I (a dose-escalation part) will explore multiple dose levels, pharmacokinetics (PK), and select a single dose level to explore in Phase II of the study. A conventional 3+3 design will be utilized. Once a dose level is selected, an additional cohort of 3-6 patients will be enrolled to assess more effectively the safety during 2 treatment cycles and confirm Phase II dose (P2D).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- KLS-1 dose escalation Phase I - Cohort 1: 2.0 mg/kg (Experimental): 3-6 patients will receive KLS-1 at 2.0 mg/kg.
  Interventions: Drug: Zinc-64 Aspartate
- KLS-1 dose escalation Phase I - Cohort 2: 3.0 mg/kg (Experimental): 3-6 patients will receive KLS-1 at 3.0 mg/kg.
  Interventions: Drug: Zinc-64 Aspartate
- KLS-1 dose escalation Phase I - Cohort 3: 3.9 mg/kg (Experimental): 3-6 patients will receive KLS-1 at 3.9 mg/kg.
  Interventions: Drug: Zinc-64 Aspartate
- KLS-1 dose escalation Phase I - Cohort 4: 4.75 mg/kg (Experimental): 3-6 patients will receive KLS-1 at 4.75 mg/kg.
  Interventions: Drug: Zinc-64 Aspartate
- KLS-1 dose escalation Phase I - Cohort 5: 6.5 mg/kg (Experimental): 3-6 patients will receive KLS-1 at 6.5 mg/kg.
  Interventions: Drug: Zinc-64 Aspartate
- KLS-1 dose expansion Phase II cohort (Experimental): The Phase II dose (P2D) defined in Phase I will be administered in a dose expansion cohort during 5 weeks of continuous bi-weekly administration of KLS-1, demonstrating that this dose was well-tolerated and safe.
  Interventions: Drug: Zinc-64 Aspartate

INTERVENTIONS:
Drug: Zinc-64 Aspartate — KLS-1 drug substance is Zinc Aspartate enriched with isotope Zinc-64 to 99.2% mass fraction of total Zinc. KLS-1 investigational medicinal product (IMP) is formulated as a solution, containing 25.64 mg of drug substance in 1 ml and inactive ingredients (water for injections, USP, EuPh).
  Other Names: KLS-1

SUMMARY:
The goal of this clinical trial is to test the safety and preliminary efficacy of a new drug, KLS-1, in adults with different types of solid tumors and chronic lymphocytic leukemia (CLL). The main questions it aims to answer are:

* To define Dose Limiting Toxicities (DLT) and maximum tolerated dose (MTD) of KLS-1
* To select the recommended Phase II Dose (P2D) of KLS-1
* To determine the single dose and multiple dose PK profile following IV administration of KLS-1
* What is the safest and most effective dose of KLS-1?
* Does KLS-1 show anti-tumor activity in patients?
* To evaluate preliminary efficacy of KLS-1 in up to 4 cohorts of locally advanced or metastatic solid tumor (malignant melanoma, prostate cancer, pancreatic cancer), or CLL.
* To evaluate 12-months progression-free survival (PFS) and duration of response (DOR) follow-up after the last dose of KLS-1

Participants will:

* Receive KLS-1 through intravenous (IV) infusions in 21-day cycles.
* Be monitored for side effects and improvements in their malignancy. Investigators will compare different doses of KLS-1 in the initial phase to find the best dose for Phase II. Once the P2D is defined, it will be tested in a larger group to see its effects on locally advanced or metastatic solid tumor (malignant melanoma, prostate cancer, pancreatic cancer) and CLL.

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, non-randomized, multicenter study of KLS-1 administered via intravenous (IV) infusions in 21-day treatment cycles to adult participants with different types of solid tumors and CLL.

Phase I (a dose-escalation part) will explore multiple-dose levels, PK and select a single dose level to explore in Phase II of the study. A conventional 3+3 design will be utilized. Once a dose level is selected, the additional cohort of 3-6 patients will be enrolled to assess more effectively the safety during 2 treatment cycles and confirm Phase II dose (P2D). Phase II (a dose expansion part) will evaluate the evidence of anti-tumor activity of the selected dose in four dose expansion cohorts of patients with different types of solid locally advanced and/or metastatic tumors or CLL. The study is designed to identify and characterize the safety, tolerability, efficacy, and PK profile of KLS-1 in oncological patients.

ELIGIBILITY:
Inclusion Criteria:

Phase I and Phase II - solid tumors cohorts

1. Adult (male or female) aged ≥18 years.
2. Signed informed consent prior to any study-specific procedures.
3. Patients who are willing to make themselves available for the duration of the study and are willing to follow study procedures.
4. Have a performance status on the Eastern Cooperative Oncology Group (ECOG) scale of:

   Phase I - 0 or 1; Phase II - 0-2.
5. Have an estimated life expectancy of ≥12 weeks.
6. Have adequate organ function including:

   a. Hematologic:
   * ANC ≥1.5 x 109/L
   * Platelets ≥100 x 109/L
   * Hemoglobin ≥90 g/L b. Hepatic:
   * Albumin ≥30 g/L
   * Bilirubin ≤1.5 times upper limit of normal (ULN)
   * ALT and AST ≤2.5 x ULN. If the liver has tumor involvement, AST and ALT ≤5 x ULN are acceptable.

     c. Renal:
   * Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 d. Blood coagulation:
   * International Normalized Ratio (INR) or activated partial prothrombin time (aPTT) <1.5 x ULN and > 0.8 x LLN lower limit of normal (LLN).
7. Have discontinued all chemotherapy, investigational therapy, molecularly targeted therapy, and cancer-related hormonal therapy at least 30 days prior to study enrollment (6 weeks for mitomycin-C or nitrosoureas).
8. Have discontinued biologic therapy and immunotherapy at least 21 days prior to study enrollment.
9. Patients who have had radiation therapy must be fully recovered in the opinion of the investigator prior to enrolling on study.
10. Are recovered or recovering from the acute adverse effects of any chemotherapy, biologic therapy, immunotherapy, molecularly-targeted therapy, cancer-related hormonal therapy, and investigational therapy (≤Grade 1 or baseline), with the exception of alopecia or Grade 2 neuropathy.
11. Have received at least 1 but no more than 4 prior systemic therapies for CLL.
12. Patients who have had surgery must be fully recovered in the opinion of the investigator prior to enrolling on study (but not less than 28 days for major surgery and 14 days for minor surgery).
13. Female patients with reproductive potential must agree to use 2 forms of highly effective contraception during the study and for at least 3 months following the last dose of IMP. Sexually active male patients must use a barrier method of contraception (condom) during the study and for at least 3 months following the last dose of IMP.
14. Females with child-bearing potential must have had a negative pregnancy test result ≤28 days prior to the first dose of IMP, as well as ≤1 day prior to the first dose of IMP.
15. Patients must be, in the judgment of the investigator, appropriate candidates for experimental therapy, and no standard therapy would confer clinical benefit to the patients.
16. Patients must have at least one lesion that is measurable by RECIST v.1.1.

Phase I 17. Patients must have histologically proven evidence of any type of metastatic solid tumor (excluding primary brain tumor) that is evaluable and for whom no approved therapy with demonstrated clinical benefit is available or patients who are intolerant or have declined standard therapy.

Phase II 18. Patients must have histologically proven evidence of a solid tumor that is locally advanced and/or metastatic and for whom no approved therapy with demonstrated clinical benefit is available or patients who are intolerant or have declined standard therapy as follows:

1. Cutaneous melanoma
2. Prostate cancer
3. Pancreatic cancer

Phase II - CLL cohort

1. Adult (male or female) aged ≥18 years.
2. Signed informed consent prior to any study-specific procedures.
3. Patients who are willing to make themselves available for the duration of the study and are willing to follow study procedures.
4. Subjects with confirmed diagnosis of per iwCLL 2008.
5. Documented disease progression that meets at least one of the iwCLL criteria for requiring treatment.
6. Measurable disease defined by either absolute lymphocyte count (ALC ≥ 5 x 109/L) or nodal lesion by computed tomography (CT).
7. Have a performance status on the Eastern Cooperative Oncology Group (ECOG) scale ≤ 2.
8. Have an estimated life expectancy of ≥16 weeks.
9. Have adequate organ function including:

   a. Adequate hematologic function in the absence of transfusions (within 6 weeks prior to first dose of study medication) and independent of growth factor support for at least 7 days with the exception of pegylated G-CSF which requires at least 14 days, defined as:
   * WBC ≥3.0 x 109/L
   * ANC ≥1.0 x 109/L
   * Platelets ≥50 x 109/L or ≥ 25 × 109/L if thrombocytopenia is related to CLL b. Hepatic:
   * Albumin ≥30 g/L
   * Bilirubin ≤2 x ULN. Subjects with known Gilbert's Syndrome or disease-related hemolysis must have a total bilirubin ≤ 3 x ULN
   * ALT and AST ≤2.5 x ULN. c. Renal:
   * Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 d. Blood coagulation:
   * International Normalized Ratio (INR) or activated partial prothrombin time (aPTT) <1.5 x ULN and > 0.8 x LLN.
10. Have discontinued all chemotherapy, immunotherapy, investigational therapy, biologic therapy, molecularly targeted therapy, and cancer-related hormonal therapy at least 30 days prior to study enrollment (6 weeks for mitomycin-C or nitrosoureas).
11. Are recovered or recovering from the acute adverse effects of any chemotherapy, biologic therapy, immunotherapy, molecularly targeted therapy, cancer-related hormonal therapy, and investigational therapy (≤Grade 1 or baseline), with the exception of alopecia or Grade 2 neuropathy.
12. The subject must also agree to pretreatment and on-treatment bone marrow aspirates.
13. Have received at least 1, but not more than 3 prior lines of therapy according to current guidelines.
14. Patients who have had surgery must be fully recovered in the opinion of the investigator prior to enrolling on study (but not less than 28 days for major surgery and 14 days for minor surgery).
15. Female patients with reproductive potential must agree to use 2 forms of highly effective contraception during the study and for at least 3 months following the last dose of IMP. Sexually active male patients must use a barrier method of contraception (condom) during the study and for at least 3 months following the last dose of IMP.
16. Females with child-bearing potential must have had a negative pregnancy test result ≤28 days prior to the first dose of IMP, as well as ≤1 day prior to the first dose of IMP.
17. Patients must be, in the judgment of the investigator, appropriate candidates for experimental therapy, and no standard therapy would confer clinical benefit to the patients.

Exclusion Criteria:

1. Have another tumor of another location except basal cell carcinoma.
2. Have a history of organ transplant (e.g., heart, lungs, liver, bone marrow, or kidney).
3. Females who are pregnant or breastfeeding.
4. Have symptomatic human immunodeficiency virus (HIV) infection, known HIV positive test results or have chronic active hepatitis B or C (screening is not required).
5. Positive COVID-19 test or signs of coronavirus infections.
6. Have clinically significant cardiac disease including any of the following:

   * A history of congenital long QT syndrome, symptomatic bradycardia, ventricular arrhythmia, uncontrolled atrial fibrillation, second- or third-degree heart block, or other conduction abnormality that in the opinion of the investigator would preclude safe participation in this study.
   * Congestive heart failure (New York Heart Association Class ≥3).
   * Unstable angina pectoris, acute myocardial infarction, or stroke ≤12 months prior to enrollment.
   * QTcF prolongation >450 msec.
7. Currently taking medication known to prolong the QT interval or induce TdP, which cannot be discontinued or substituted.
8. Uncontrolled type 1 or 2 diabetes with high risk of hypoglycemia.
9. Are a family member of the investigator or staff of the study site.
10. Are currently enrolled in another interventional clinical study of an investigational therapy.
11. Hypersensitivity to any components of KLS-1. Additional exclusion criterion for patients enrolled in Phase II to CLL cohort
12. History of Richter's transformation or prolymphocytic leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Cycle 1 Day 1, Cycle 1 Day 3, Cycle 1 Day 6, Cycle 1 Day 9, Cycle 1 Day 12, Cycle 1 Day 21, 30-Day Follow-Up (Each cycle is 28 days)
  Dose Limiting Toxicities (DLTs) at Dose Escalation Cohorts
Number of participants with Dose Limiting Toxicities (DLTs) | Cycle 1 Day 1, Cycle 1 Day 3, Cycle 1 Day 6, Cycle 1 Day 9, Cycle 1 Day 12, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 6, Cycle 2 Day 12, Cycle 2 Day 21, 30-Day Follow-Up (Each cycle is 28 days)
  Dose Limiting Toxicities (DLTs) at Dose Confirmation Cohorts
Number of participants with Treatment Emergent Adverse Events (AEs) | Cycle 1 Day 1, Cycle 1 Day 3, Cycle 1 Day 6, Cycle 1 Day 9, Cycle 1 Day 12, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 6, Cycle 2 Day 12, Cycle 2 Day 21, 30-Day Follow-Up (Each cycle is 28 days)
  Adverse Events (AEs) as characterized by type, frequency, severity as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, timing, seriousness and relationship to study therapy
Number of participants with Treatment Emergent Serious Adverse Events (SAEs) | Cycle 1 Day 1, Cycle 1 Day 3, Cycle 1 Day 6, Cycle 1 Day 9, Cycle 1 Day 12, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 6, Cycle 2 Day 12, Cycle 2 Day 21, 30-Day Follow-Up (Each cycle is 28 days)
  Serious Adverse Events (SAEs) as characterized by type, frequency, severity as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, timing, seriousness and relationship to study therapy
Number of participants with Overall Response Rate (ORR) | 30-Day Follow-up, Q 3-Months Follow-up, 12-Months Follow -up
  ORR evaluated upon using RECIST, version 1.1 and the based on International Workshop on Chronic Lymphocytic Leukemia (iwCLL) response criteria per Investigator assessment

SECONDARY OUTCOMES:
Cmax of KLS-1 | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: maximum plasma concentration (Cmax) of KLS-1
AUC0-t and AUC0-∞ of KLS-1 | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: area under the plasma concentration-time curve (AUC0-t and AUC0-∞) of KLS-1
T1/2 of KLS-1 | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: Half-Life (T1/2) of KLS-1
Tmax of KLS-1 | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: time to reach maximum plasma concentration (Tmax) of KLS-1
CL/F of KLS-1 | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: clearance (CL/F) of KLS-1
Vd/F of KLS-1 | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: apparent volume of distribution (Vd/F) of KLS-1
Ae(0-t) of Zinc | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: cumulative amount of Zinc excreted in urine (Ae(0-t))
Rmax of Zinc | Cycle 1 Day 1,Cycle 1 Day 3, Cycle 1 Day 9, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 3, Cycle 2 Day 21 (Each cycle is 28 days)
  PK parameters: maximum ate of urinary excretion (Rmax) of Zinc

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Valerii Cheshuk, MD, PhD, Principal Investigator — Medical Centre of Arensia Exploratory Medicine LLC
Locations (1):
- Medical Centre of Arensia Exploratory Medicine LLC, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No